CLINICAL TRIAL: NCT04596124
Title: Clincal Evaluation of the Effectiveness and Tolerability of Fitostimoline Plus Cream and Fitostimoline Plus Gauze vs Connettivina Bio Plus Cream and Connettivina Bio Plus Gauze in the Treatment of Acute Skin Lesions
Brief Title: Effectiveness and Tolerability of Fitostimoline Plus Cream and Gauze vs Connettivina Bio Plus Cream and Gauze
Acronym: FP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Farmaceutici Damor Spa (Industry)
Responsible Party: Principal Investigator, carmine alfano, PROFESSOR, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fitostimoline plus
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Wound Heal; Wound Infection; Wounds and Injuries
MeSH Terms: conditions — Wound Infection; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: randomized, controlled, multicentric study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- fitostimoline plus cream (Experimental)
  Interventions: Device: fitostimoline plus
- fitostimoline plus gauze (Experimental)
  Interventions: Device: fitostimoline plus
- connettivina bio plus cream (Active Comparator)
  Interventions: Device: fitostimoline plus
- connettivina bio plus gauze (Active Comparator)
  Interventions: Device: fitostimoline plus

INTERVENTIONS:
Device: fitostimoline plus — randomized controlled multicentric study
  Other Names: connettivina bio plus

SUMMARY:
This study aims to compare the efficacy and clinical tolerability of two medical devices in gauze and cream containing the aqueous extract of triticum vulgare and polyhexanide in comparison with two medical devices containing hyaluronic acid and silver sulfadiazine in the treatment of acute skin lesions . The reason why the two types of devices are compared is because hyaluronic acid and silver sulfadiazine represent the gold standard for the treatment of acute skin lesions. Therefore, making a comparison between the activity of the aqueous extract of triticum vulgare and polyhexanide and this gold standard of control in the treatment of acute skin lesions, is useful to better define the efficacy and tolerability of both medical devices in order to eventually expand the therapeutic armamentarium available for the treatment of acute skin lesions

DETAILED DESCRIPTION:
Skin lesions, more or less deep, are areas of rupture and tissue loss with exposure of the underlying tissues.

The term "external lesion" or "wound" indicates the morphological and functional destruction of the continuity of the superficial skin layers and, in the most serious cases, of the deep subcutaneous layers.

The lesions are evaluated and cataloged on the basis of their width, depth and characteristics. Furthermore, the development, the causes (etiopathogenesis) and the pathophysiological context of the wound are considered.

Superficial, slight lesions affect only the epidermis, the dermis and at most part of the hypodermis; the deeper ones involve all the subcutaneous tissue (fat) up to the muscles, the periosteum, reaching the exposure of the bone or supporting structures (tendons and cartilages); the most severe (chronic) are characterized by loss of substance in the skin and a poor tendency to healing.

According to the timing of healing, the lesions are divided into acute and chronic.

Acute injuries heal through 3 different phases and reach tissue repair within 8/10 weeks. Beyond this time the lesion becomes chronic and, if not acted correctly, the wound becomes more complicated and degrades in increasingly serious stages / degrees.

The acute wounds that the healthcare professional must treat most frequently are surgical wounds. Depending on their extent, acute wounds can be distinguished into stab wounds, puncture wounds, lacerated wounds and lacerated-contused wounds.

This type of acute wounds can generally heal in a physiological way or be induced to healing through the use of dressings, which reduce healing times.

The main dressings used to treat these lesions are hyaluronic acid-based dressings containing antiseptics, such as silver sulphadiazine to prevent the risk of contamination and colonization by microorganisms. In these dressings, hyaluronic acid promotes the acceleration of the tissue repair process.

However, among the main products used by hospital and non-hospital surgeries there are also dressings based on Rigenase® (aqueous extract of triticum vulgare) and polyhexanide. Rigenase®, containing the aqueous extract of triticum vulgare, has pro-proliferative, anti-inflammatory and antioxidant activity. These activities are attested by recent literature which indicates that the aqueous extract of triticum vulgare has pro-proliferative activity on fibroblasts and keratinocytes, the main cells involved in proliferation during the lesion repair process; in addition, the aqueous extract of triticum vulgare also has a documented anti-inflammatory activity, mediated by the reduction of the main cytokines responsible for skin inflammation, and an anti-metalloprotease9 activity, the main actor of inflammation in skin lesions. The antioxidant activity of Rigenase®, verified on the hemolysis of erythrocytes, is comparable to that of ascorbic acid.

The activity of polyhexanide is also fundamental for the prevention of the risk of colonization and contamination by microorganisms in acute skin lesions. In fact, this latest generation antiseptic has a consolidated antiseptic activity on gram positive and gram negative bacteria, on fungi and on some viruses, without the development of resistance both in vitro and in vivo.

Based on the foregoing, this study aims to compare the efficacy and clinical tolerability of two medical devices in gauze and cream containing the aqueous extract of triticum vulgare and polyhexanide in comparison with two medical devices containing hyaluronic acid and silver sulfadiazine. in the treatment of acute skin lesions. The reason why the two types of devices are compared is because hyaluronic acid and silver sulfadiazine represent the gold standard for the treatment of acute skin lesions. Therefore, making a comparison between the activity of the aqueous extract of triticum vulgare and polyhexanide and this gold standard of control in the treatment of acute skin lesions, is useful to better define the efficacy and tolerability of both medical devices in order to to possibly expand the therapeutic armamentarium available for the treatment of acute skin lesions

ELIGIBILITY:
Inclusion Criteria:

* Outpatient patients (regardless of sex) aged 18 and over;
* Presence of acute injury
* Willingness to cooperate and ability to understand the procedures and purposes of the study;
* Willingness to take part in the study and to adhere to the experimental procedures certified by signing the written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Inadequate contraceptive procedures in fertile women;
* Anamnestic data of any local and / or systemic pathology potentially able to interfere with the study parameters;
* Chronic concomitant treatment with local antiseptics, anti-inflammatory drugs (steroid and non-steroidal), analgesic, antineoplastic, immunosuppressive drugs;
* Immunodeficiency states (eg HIV infection); neoplastic diseases in progress;
* Non-therapeutic use of psychoactive substances;
* Abuse of drugs and / or alcohol;
* Neurological disorders or psychiatric conditions that may affect the validity of the consent and / or compromise the patient's adherence to the study procedures;
* Allergy, hypersensitivity or intolerance known to the constituents of the preparations under study;
* Any condition, medical or otherwise, that could significantly reduce the possibility of obtaining reliable data, achieve the objectives of the study, refine the completion of this;
* Presumption of poor reliability or collaboration;
* Treatment with any investigational drug in the last 30 days prior to the start of the study;
* Patients already enrolled in this study;
* Center staff directly involved in the management of the study and close relatives of that.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-08-18 (Estimated); Study Completion 2022-09-18 (Estimated)

PRIMARY OUTCOMES:
Total symptom score | 46 days
  Total symptom score will be measured by a scale from 0 (absence of symptoms) to 4 (maximum intensity of symptoms).

SECONDARY OUTCOMES:
Visual Analog Scale | 46 days
  The visual analog scale will be evaluated for the presence of subjective acute and chronic pain. Scores will be recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: carmine alfano, Principal Investigator — università di salerno
Locations (1):
- Barbara Maglione, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No